CLINICAL TRIAL: NCT00596518
Title: A Phase 1, Open-Label Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of PF-00734200 Administered To Subjects With Various Degrees Of Renal Impairment And Normal Renal Function
Brief Title: A Study to Evaluate the Blood Levels, Safety, and Tolerability of PF-00734200 in Subjects With Impaired Kidney Function and Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A7941014
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — gosogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-00734200 (Experimental)
  Interventions: Drug: PF-00734200

INTERVENTIONS:
Drug: PF-00734200 — The drug is administered as a single dose of four 5-mg tablets

SUMMARY:
The purpose of this study is to compare how PF-00734200 is adsorbed, distributed, broken down and eliminated by subjects with mild, moderate and severe kidney impairment, by subjects receiving chronic hemodialysis, and by subjects with normal kidney function. The removal rate of PF-00734200 by hemodialysis will be calculated. The safety and tolerability of PF-00734200 in subjects with various degrees of kidney function or undergoing chronic hemodialysis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet one of the following renal function categories Normal renal function Mild renal impairment Moderate renal impairment End stage renal disease requiring chronic hemodialysis
2. Body mass index between approximately 18-40 kg/m2 inclusive, and a total body weight greater than 50 kg
3. Subjects in the normal renal function category must be healthy and not receiving any chronic treatment with prescription or non-prescription medications

Exclusion Criteria:

1. Women who are pregnant, nursing or women of childbearing potential
2. Subjects with acute renal disease.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 until last observation (AUCtlast) | 3-6 days
Maximum serum concentration (Cmax) | 3-6 days

SECONDARY OUTCOMES:
AUC extrapolated to infinity (AUCinf) | 3-6 days
Time of Cmax (Tmax) | 3-6 days
Half life (T1/2) | 3-6 days
Renal clearance (CLr) | 3-6 days
Hemodialysis clearance (CLd) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Knoxville, Tennessee